CLINICAL TRIAL: NCT03005574
Title: A Randomized Controlled Trial Comparing the Impact of Thinking Skills for Work (TSW)Tablet-based Home Practice Program on Cognitive Functioning and Work With the Traditional TSW Program
Brief Title: Comparing Thinking Skills for Work (TSW)Home Practice Program With Traditional TSW Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Susan Mcgurk, Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4391
Record Dates: First submitted 2016-12-26; First posted 2016-12-29 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Major Depression
Keywords: Severe Mental Illness; Cognitive Remediation; Employment
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TSW-HP (Experimental): TSW-HP Intervention implemented by a cognitive specialist over a 6-month treatment period which includes 24 hours (1 hour per week) of facilitated cognitive exercise sessions, which will be supplemented by approximately 24 hours of home practice sessions on a tablet computer.
  Interventions: Behavioral: TSW-HP
- TSW-T (Active Comparator): Participants assigned to traditional TSW will receive the usual TSW program, which includes a one hour cognitive exercise practice session per week at Brooklyn Community Services (BCS) for 6 months. This group will not receive home based cognitive practice exercises.
  Interventions: Behavioral: TSW-T

INTERVENTIONS:
Behavioral: TSW-HP — TSW-HP involves home practice of cognitive exercises along with the training sessions facilitated by the cognitive specialist at the agency.
  Arms: TSW-HP
Behavioral: TSW-T — Participants assigned to traditional TSW will receive the usual TSW program which includes a one hour session per week at BCS for 6 months. This group will not receive home based cognitive practice exercises
  Arms: TSW-T

SUMMARY:
The purpose of this study is to determine if using a tablet computer, which is a very small, easy-to-carry computer, to practice thinking exercises at home will help improve your attention, memory, and problem solving abilities. All the participants will receive training in the thinking skills for work program. But in order to determine the effect of tablet use for home practice, half of the participants will be given a tablet to practice the thinking exercises at home. All participants will be receiving vocational rehabilitation and have a goal of getting a job.

DETAILED DESCRIPTION:
The Thinking Skills for Work (TSW) program has been shown to improve cognitive functioning and work in multiple studies in a variety of vocational programs. TSW includes agency-based, computer cognitive practice facilitated by a cognitive specialist, and teaching of compensatory strategies to manage cognitive challenges, which are integrated with vocational services. Supplementing agency-based practice with home practice on a tablet addresses the need and desire for more cognitive practice, which is expected to further improve cognitive and work outcomes.

This randomized controlled trial will evaluate the impact of supplementing the traditional TSW cognitive practice with home based practice of cognitive exercises using a tablet.. Fifty clients enrolled in vocational services at Brooklyn Community Services will be recruited and randomized either to TSW-Home Practice (N=25) or traditional TSW (N=25).

All the participants will be assessed at baseline, 6 months and 12 months on cognitive functioning and symptoms; work activity will be tracked for 12 months; program satisfaction will be assessed at 6 and 12 months. The study will establish the efficacy of using home practice on a tablet to increase the number of computer cognitive practice exercises completed by clients.

Study hypotheses: 1) Individuals assigned to TSW HP will complete more cognitive practice sessions using COGPACK software than those assigned to traditional TSW; 2) Individuals who are exposed to TSW HP (i.e., complete 6 or more cognitive practice sessions) will complete more practice sessions than those who are exposed to traditional TSW; 3) Individuals assigned to TSW - HP will show greater improvements in cognitive functioning at post treatment and follow up than those assigned to traditional TSW; 4) Individuals assigned to TSW - HP will show greater improvements in work related outcomes (number of job interviews, % obtaining competitive work, weeks worked, wages earned) at post-treatment and follow up than those assigned to traditional TSW.

ELIGIBILITY:
Inclusion Criteria:

age 18 years or older; severe mental illness based on New York State Office of Mental Health criteria; not competitively employed but want to work; enrolled in vocational rehabilitation at Brooklyn Community Services; fluent in English.

Exclusion Criteria:

prior receipt of more than 3 sessions of Thinking Skills for Work (TSW) Cognitive Remediation; medical disorder with known effects on cognitive functioning; inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Composite Measure of Change in Neurocognitive Functioning | 6 months and 12 months
  Neurocognitive tests for primary outcome variables are from (MATRICS) Consensus Cognitive Battery

CONTACTS AND LOCATIONS:
Overall Officials: Susan R McGurk, PhD, Principal Investigator — Boston University
Locations (1):
- Brooklyn Community Services, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No